CLINICAL TRIAL: NCT02737397
Title: A Double-blind Placebo-controlled 4-Way Crossover Study to Evaluate the Efficacy of JMI-001 (an Over-the-counter Pain Medicine and an Antihistamine) in the Prophylaxis of Veisalgia in Healthy Volunteers
Brief Title: Safety and Efficacy of a Combination Product for the Prevention of Veisalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sen-Jam Pharmaceutical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: JMI-001-001
Record Dates: First submitted 2016-03-22; First posted 2016-04-13 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Veisalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- pain medicine and antihistamine (Experimental): JMI-001 (SJP-304 and SJP-223)
  Interventions: Drug: JMI-001 (SJP-304 and SJP-223)
- pain medicine (Active Comparator): SJP-304 and placebo
  Interventions: Drug: SJP-304; Drug: placebo
- antihistamine (Active Comparator): SJP-223 and placebo
  Interventions: Drug: SJP-223; Drug: placebo
- placebo (Placebo Comparator): placebo and placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: JMI-001 (SJP-304 and SJP-223)
  Arms: pain medicine and antihistamine
Drug: SJP-304
  Arms: pain medicine
Drug: SJP-223
  Arms: antihistamine
Drug: placebo
  Arms: antihistamine; pain medicine; placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a combination product for the prevention of veisalgia. Common symptoms of veisalgia following the moderate consumption of alcohol includes headache, fatigue, and thirst. It is the investigators hypothesis that a combination of two drugs can alleviate or significantly reduce these symptoms when taken before the start of moderate alcohol consumption.

DETAILED DESCRIPTION:
Some people who consume alcohol in moderation experience veisalgia. These symptoms include a long list of adverse effects that include headache, fatigue and thirst. The mechanism by which these effects occur has not been fully elucidated. Although, it has been documented that alcohol causes the release of a large number of substances into the blood stream that cause a number of physiologic changes.

A 4-arm study will help to determine the effect each agent contributes to decreasing the alcohol induces physiologic changes and the effect when the two agents are delivered concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonsmoking men or women between 25 and 65 years inclusive
* Good general health as determined by a thorough medical history and physical examination including vital signs
* Subject is a self-reported moderate drinker of alcohol. Moderate drinking can be approximated with a blood alcohol concentration (BAC) of 0.04 - 0.11%. The 0.04% - 0.11% BAC correlates approximately with a 120-160 pound female drinking 2 to 5 drinks in 2 to 3 hours, respectively, and a 160-200 pound male drinking 3 to 7 drinks in 2 to 3 hours, respectively.
* Subject has had a moderate to heavy drinking episode in the past 90 days that produced hangover symptoms
* Subject is knowledgeable of the amount of alcohol he/she needs to consume over a 2 to 3 hour period of time to produce hangover symptoms
* Body mass index between 19 and 32 kg/m2, inclusive
* Report a regular, habitual bedtime between 21:30 and 24:00
* Females of childbearing potential must be using an acceptable method of contraception (see Section 8.5) or have been surgically sterilized and have a negative urine pregnancy test at screening and upon admission for each treatment visit
* Subject is capable of understanding the requirements of the study and to give written informed consent
* Subject is able to follow study instructions and is willing to complete all study visits and procedures

Exclusion Criteria:

* Acute illness within 14 days prior to screening visit
* Allergic reaction or upper respiratory tract infection within 7 days of screening visit
* Vaccination administration within 7 days of screening visit
* Clinically significant, unstable medical illness
* Evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic or neurological disease
* History of cancer or diabetes
* Subject has a previous or current Substance-Related Disorder as defined by DSM-5
* Self-report of a usual consumption of more than 14 units of alcohol per week. One unit of alcohol is equivalent to 12 ounces of beer, 4 ounces of wine, or

  1 ounce of liquor
* Self-report of recent (within one month) or current use of smoked or chewed tobacco products, or use of nicotine (e.g., nicotine gum or patch)
* Positive alcohol breathalyzer test at screening or at check-in for any treatment visit
* Positive urine drug screen at screening or at check-in for any treatment visit
* A supine blood pressure > 140/90 mm/Hg at screening
* Heart rate > 100 beats per minute at screening
* Subjects who are unwilling to forgo caffeine consumption with or following dinner on each treatment night or who are unwilling to comply with study restrictions for prohibited medications/ foods throughout study participation.
* Clinically significant psychiatric illness, including chronic psychiatric illness or the history or presence of any Axis I condition
* Any clinically significant abnormal finding on physical examination or vital signs
* Positive pregnancy test at screening or at check-in for any treatment visit
* Subject has previously experienced an allergic reaction or adverse event associated with aspirin, NSAIDs, or antihistamine usage, including a reaction of not effective
* Subject is taking any prescription or over-the-counter oral pain medication(s) for any reason
* Subject is taking prescription or over-the-counter antihistamine(s)
* Women who are pregnant or breastfeeding
* Any medical condition or any condition or situation that in the investigator's opinion may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study
* Concurrent participation in an investigational drug or device study, or use of any investigational drug within 30 days prior to screening

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magdy L Shenouda, Principal Investigator — Clinilabs, Inc.

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 4 way cross-over study where 13 individuals received a single dose of an agent in a randomized sequence. All participants were intended to receive all four interventions.
Groups:
- All Study Participants: JMI-001 (SJP-304 and SJP-223), single dose
  SJP-304 + placebo
  SJP-223 + placebo
  placebo + placebo
Period: Overall Study
Arm/Group | All Study Participants
Started | 13
JMI-001 | 13
SJP-304 | 12
SJP-223 | 13
Placebo | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomized to receive 4 sequences of drug therapy including placebo.
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Veisalgia with pre-determined consumption [Count of Participants; unit: Participants] | 13

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Side Effect Prevention Using the Acute Hangover Scale
Description: Efficacy of pain medicine + antihistamine in reducing (as compared to placebo) symptoms associated with Veisalgia. The Acute Hangover Scale (AHS) will be used to evaluate side effects on the following morning post alcohol consumption. The scale includes 9 symptom assessments each ranging from 0-10. The total score can range from 0-90. (0= no symptoms, 10 = worst symptom ever).
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pain Medicine: SJP-304 and placebo
  SJP-304
  placebo
- Antihistamine: SJP-223 and placebo
  SJP-223
  placebo
- Placebo: Placebo + placebo, single dose
Arm/Group | Pain Medicine and Antihistamine | Pain Medicine | Antihistamine | Placebo
Number analyzed (Participants) | 13 | 12 | 13 | 13
score on a scale | 6.7 (5.66) | 4.7 (5.05) | 7.8 (8.66) | 6.8 (7.21)

2. Post Hoc Outcome: Efficacy of Side Effect Prevention Using the Acute Hangover Scale (Hangover Sensitive Subpopulation)
Description: as for outcome 1
Time Frame: 24 hours
Population: A subset of participants were analyzed post-hoc that were hangover sensitive when compared to placebo.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Medicine and Antihistamine | Pain Medicine | Antihistamine | Placebo
Number analyzed (Participants) | 5 | 4 | 5 | 5
score on a scale | 7 (4.1) | 6 (6.5) | 9 (6.9) | 13.4 (7.7)

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Placebo: placebo and placebo
  placebo
Arm/Group | Pain Medicine and Antihistamine | Pain Medicine | Antihistamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 0/12 | 0/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pain Medicine and Antihistamine (N=13) | Pain Medicine (N=12) | Antihistamine (N=13) | Placebo (N=13)
epigastric pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — treatment not necessary

LIMITATIONS AND CAVEATS:
Participants were not tested and excluded for hangover insensitivity, prior to being entered into the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No